CLINICAL TRIAL: NCT02286622
Title: A Single Dose Evaluation of the Effects of Renal Impairment on Deflazacort Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MP-104-CL-024
Record Dates: First submitted 2014-11-04; First posted 2014-11-10 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — deflazacort

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Renal Impairment (Experimental): Eight (8) subjects with ESRD on HD will receive one 18 mg dose of deflazacort.
  Interventions: Drug: Deflazacort
- Healthy Volunteers (Experimental): Eight (8) healthy subjects with estimated creatinine clearance (CLcr) ≥ 90 mL/min. Subjects will be matched for age [± 15 years], BMI [± 15 %], and gender [1:1] to the subjects in the ESRD cohort. Subjects will receive one 18 mg dose of deflazacort.
  Interventions: Drug: Deflazacort

INTERVENTIONS:
Drug: Deflazacort — Deflazacort, a glucocorticoid with anti-inflammatory and immunosuppressive effects, is used in treating a variety of diseases. Pharmacologically it is an inactive pro-drug which is metabolized immediately to the active metabolite 21-desacetyl-DFZ. The elimination of this metabolite is primarily via the urine in humans. Its potency is approximately 70 to 90% of prednisone and 6 mg of deflazacort has approximately the same anti-inflammatory potency as 5 mg of prednisolone or prednisone
  Other Names: DFZ

SUMMARY:
This is a non-randomized, open-label, single-dose study to compare the PK of 21 desacetyl-DFZ and, if data permits, deflazacort in 8 subjects with ESRD to that of 8 healthy matched control subjects (age, body mass index [BMI], and gender).

DETAILED DESCRIPTION:
This is a non-randomized, open-label, single-dose study to compare the PK of 21 desacetyl-DFZ and, if data permits, deflazacort in 8 subjects with ESRD to that of 8 healthy matched control subjects (age, body mass index [BMI], and gender).

All subjects with ESRD will be on hemodialysis (HD). Dosing of deflazacort followed by PK evaluation of 21 desacetyl DFZ and, if data permits, deflazacort, will only be performed on a non-HD day.

On Day 1, that will be scheduled on a non-HD day for subjects with ESRD, a single oral dose of deflazacort will be administered followed by serial blood sampling for 24 hours to assess the PK of 21 desacetyl-DFZ, and, if data permits, deflazacort.

Safety will be monitored throughout the study by repeated clinical and laboratory evaluations.

Subjects will return to the Clinical Research Unit (CRU) 3 days (± 1 day) following study drug administration to determine if any adverse events (AEs) have occurred since the last study visit. Subjects who terminate the study early will be contacted if the Principal Investigator (PI) deems necessary.

A total of sixteen (16) adult male and female subjects will be enrolled. Renal Impaired Cohort: Eight (8) subjects with ESRD on HD. Healthy Match Control Cohort: Eight (8) healthy subjects with estimated creatinine clearance (CLcr) ≥ 90 mL/min. Subjects will be matched for age [± 15 years], BMI [± 15 %], and gender [1:1] to the subjects in the ESRD cohort.

Each subject will receive a single oral dose of 18 mg (3 X 6 mg tablets) deflazacort, following an overnight fast.

Study drug will be administered orally with approximately 240 mL of water.

ELIGIBILITY:
Inclusion Criteria:

* Continuous non-smokers or moderate smokers
* For a female of non-childbearing potential: must have undergone a sterilization procedures or be postmenopausal with amenorrhea for at least 1 year prior to the first dose and FSH serum levels consistent with postmenopausal status
* A non vasectomized, male subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days
* If male, must agree not to donate sperm from dosing until 90 days Subject with ESRD on Hemodialysis
* Adult male or female, 18 80 years of age
* BMI ≥ 18.5 and ≤ 40.0 kg/m2 - Subject is maintained on a stable regimen of HD at least 3 months Healthy Subject
* Healthy adult male and female subjects will be matched 1:1 to a specific subject in the ESRD cohort based upon age, BMI, and gender [1:1]. The following criteria should be fulfilled:

  * 18 to 80 years of age. Age must be within ± 15 years of the matched subject's age in the ESRD cohort
  * BMI ≥ 18.5 and ≤ 40.0 kg/m2. BMI must be within ± 15% of the matched subject's BMI in the ESRD cohort
* Has a CLcr ≥ 90 mL/min

Exclusion Criteria:

* Subject is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study
* History or presence of hypersensitivity or idiosyncratic reaction to the study drugs or related compounds (e.g., steroids or their formulations including lactose and corn starh)
* History (within the last year prior to dosing) or presence of peptic ulcers
* History or presence of:

  * Gastritis or esophagitis, diverticulitis, ulcerative colitis (if there is probability of impending perforation), abscess or pyogenic infections, or fresh intestinal anastomosis
  * Previous corticoids-induced myopathy
  * Ocular herpes simplex
  * Symptomatic cardiomyopathy at screening
  * Immunosuppression or other contraindications for corticosteroid treatment
  * History of chronic systemic fungal or viral infections
  * Galactose intolerance, Lapp lactose deficiency, or glucose-galactose malabsorption
  * Osteoporosis
  * Myasthenia gravis
  * Epilepsy
  * Idiopathic hypocalcuria
* Seated blood pressure is less than 90/40 mmHg or greater than 170/100 mmHg
* Seated heart rate is lower than 40 bpm or higher than 99 bpm
* QTcF interval is > 500 msec
* Has received any live or live-attenuated vaccine within 30 days
* Has received any immunosuppressive agents, coal tar, and/or radiation therapies within 30 days
* Has received injectable corticoids in the 12 weeks prior to dosing or any oral form of corticoids in 30 days
* Unable to refrain from or anticipates the use of:

  * Any drug known to be moderate or strong inhibitors or inducers of cytochrome P450 (CYP) 3A or P-glycoprotein (P-gp) for 14 days or 28 days, respectively
  * Any medication or substance which cannot be discontinued at least 14 days
* Female subjects of childbearing potential
* Female subjects who are pregnant or lactating
* Positive results at screening for HIV, HBsAg or HCV
* Has been on a diet incompatible with the on study diet within 28 days
* Donation of blood or significant blood loss within 56 days
* Plasma donation within 7 days
* Participation in another clinical trial within 28 days Subject with ESRD
* Is a regular user of any medication that would significantly alter glomerular filtration rate, e.g., cimetidine
* Has presence of a renal carcinoma or acute renal disease caused by infection or drug toxicity
* History of drug abuse within the past 2 years
* Has a positive urine/breath alcohol or urine/serum/saliva drug testing Normal Renal Function
* History or presence of alcoholism or drug abuse within the past 2 years
* Positive urine drug or urine/breath alcohol results

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Renal impairment on the pharmacokinetics (PK) of deflazacort in subjects with end-stage renal disease including the area under the plasma concentration time curve, from time 0 to the last measurable non-zero concentration. | 1 day
  Renal impairment on the pharmacokinetics (PK) of deflazacort in subjects with end-stage renal disease including the area under the plasma concentration time curve, from time 0 to the last measurable non-zero concentration.

SECONDARY OUTCOMES:
Safety and tolerability of one dose of deflazacort in subjects with end stage renal disease as measured by capturing occurrence of adverse events. | 1 day
  Safety and tolerability of one dose of deflazacort in subjects with end stage renal disease as measured by capturing occurrence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Bioscience Center, Study Director — Marathon Pharmaceuticals, LLC
Locations (2):
- United States (2):
  - University of Miami Division of Clinical Pharmacology, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

REFERENCES:
- See also: Methylprednisolone effect on Dystrophin levels — https://www.researchgate.net/publication/14841539_Dystrophin-positive_myotubes_in_innervated_muscle_cultures_from_Duchenne_and_Becker_muscular_dystrophy_patients
- See also: Pharmacokinetics in patients with impaired ernal function — https://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/UCM204959.pdf
- See also: Deflazacort fefect on Laminin and Myogenic repair. — http://www.thelancet.com/journals/laneur/article/PIIS1474-4422(10)70196-4/fulltext
- See also: Treatment of DMD-Worsening of Cardiomyopathy — http://www.oalib.com/references/12905458
- See also: Deflazacort Vs Prednisone in DMD — http://onlinelibrary.wiley.com/doi/10.1002/1097-4598(200009)23:9%3C1344::AID-MUS4%3E3.0.CO;2-F/full